CLINICAL TRIAL: NCT01131819
Title: Use of an Interactive Video Game as Part of a New Amputee Rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, William C. Miller, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H09-00523
Record Dates: First submitted 2010-05-21; First posted 2010-05-27 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Below Knee Amputation
Keywords: Trans-tibial Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): The novel intervention we propose to use, the Wii Fit, will be introduced for a period of at least 20 minutes but not greater than 30 minutes per day to all the subjects in the study.
  Interventions: Device: Nintendo Wii fit ™ balance board

INTERVENTIONS:
Device: Nintendo Wii fit ™ balance board — Nintendo Wii fit ™ balance board will be introduced for a period of at least 20 minutes but not greater than 30 minutes per day to all the subjects for a minimum of 6 times in two weeks and a maximum of 18 times in 6 weeks.

SUMMARY:
Purpose: The investigators wish to determine if a rehabilitation program for subjects with new, trans-tibial amputations that has the balance portion of the program augmented by the use of the Nintendo Wii fit ™ balance board improves their performance.

Hypothesis: The investigators hypothesize that subjects will benefit from the use of the device and that this will manifest as an improvement on outcome measures.

DETAILED DESCRIPTION:
All subjects will be trained by the same specialist physiotherapist. Subjects will use the Wii Fit balance platform for a period of twenty minutes or greater per day (at the discretion of the specialist physiotherapist) during their standard rehabilitation program. These balance training exercises will be in addition to those already used in the standard rehabilitation program, but will not add to the total therapy session time. Activities on the device will be chosen by the therapist based on the subjects' current abilities and their phase of training. More complicated tasks will be given as the subject progresses. The therapist will intervene and provide instruction / correction if the subject is using unsafe technique or poor technique (postures, positioning strategies that would not be condoned in the regular training program).

The device is a stable, level platform 5.5 cm from the floor. Subjects stand on the device and may use gait aids if indicated.

Standard practice involves intensive training of the subject by the same specialist physiotherapist but without the use of the Wii Fit platform.

ELIGIBILITY:
Inclusion Criteria:

* Consented subjects with new, unilateral, transtibial amputations who are greater than 19 years of age

Exclusion Criteria:

* Subjects who have an open wound that limits their wearing of the prosthesis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery
  The Short Physical Performance Battery (SPPB) measures subject's ability to perform three tasks: standing balance, gait speed and lower extremity strength (chair stands). Collected at each data collection session
NeuroCom Clinical Research System
  The NeuroCom Clinical Research System is a commercially available objective measure that is able to detect and document perturbations in balance in three (X, Y, Z components) planes in order to determine postural sway. The system consists of a dual platform that moves or does not move in conjunction with a visual surround. The Sensory Organization Test (SOT) will be used to test 3 sensory components of balance (visual, somatosensory and vestibular inputs) under 6 standard conditions. Collected at each data collection session.

SECONDARY OUTCOMES:
Walking ability will be measured using the L-Test. This walk test incorporates a sit-to-stand component, turns to both the left and the right over a distance of 20 meters.
  Collected at each data collection session
Walking endurance will be assessed using the 2 Minute Walk Test (2MWT). Starting from a standing position this test requires individuals to walk at a fast safe pace for a period of two minutes.
  Collected at each data collection session
Balance confidence will be measured using the 16 item Activities-specific Balance Confidence (ABC Scale). The items assess the perceived confidence (self-efficacy) the individual has in performing an increasing complex series of tasks.
  Collected at each data collection session
The Short Feedback Questionnaire-modified (SFQ-M) will be used to determine subjects' level of satisfaction with their rehabilitation program as well as with the interactive video game experience.
  Collected at the end of the project
A 9-item Falls Diary will be kept by each subject documenting number of falls, circumstances (eg/ cause, location, assistive device used or not) and consequences (eg/ medical visit, injury) over the past week.
  Collected weekly

CONTACTS AND LOCATIONS:
Overall Officials: William C. Miller, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Rehab Research Lab, GF Strong Rehab Centre, Vancouver, British Columbia, Canada